CLINICAL TRIAL: NCT03799328
Title: Low Dose Multi Allergen Oral Immunotherapy for Food Allergy
Brief Title: Low Dose Multi-OIT for Food Allergy (LoMo)
Acronym: LoMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Julia Upton, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000060633
Record Dates: First submitted 2018-11-20; First posted 2019-01-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multi-OIT (Experimental): Low dose OIT with multiple allergens
  Interventions: Other: multi-OIT

INTERVENTIONS:
Other: multi-OIT — low dose OIT to multiple foods

SUMMARY:
Oral immunotherapy (OIT) is a food allergy treatment where small amounts of the food a child is allergic to is eaten and gradually increased over time with the aim to be able to eat a certain amount of the allergen without experiencing an allergic reaction. While this process works in many children there are concerns about safety, feasibility and drop-outs and how to adapt protocols for multiple allergies.

Many OIT trials have targeted approximately 4000mg of single food/day. In these trials up to 40% drop-out. There is evidence much lower doses can have beneficial effects.

The investigators will evaluate if low doses of foods can allow for OIT to multiple foods. This approach may have efficacy against accidental exposure and be able to demonstrate immune changes. This approach may have a low burden of treatment and a low rate of allergic reactions and

DETAILED DESCRIPTION:
This is a single-arm, open label, study of the intervention of low dose multiple-nut OIT in nut allergic children.

After meeting eligibility criteria, participants will have a food challenge to 2-5 nuts.

If the oral food challenge is positive, participants will be enrolled in the study to multiple nut OIT. A blood draw and quality of life (QOL) survey will occur at baseline.

Participants will have dose escalation visits of the multiple nut OIT every 2 months to a target dose of 30mg of each nut protein. A blood draw and QOL survey will occur at 6 months.

Participants will then continue with daily ingestion of the 30mg of each nut protein for 1 year with visits every 3 months.

After 18 months from the start of the study, another oral food challenge will be given to participants to assess the change in the maximum tolerated dose of nuts. A blood draw will assess changes in the immune parameters. A QOL survey will occur at 18 months to assess changes in QOL.

ELIGIBILITY:
Inclusion Criteria:

* Relevant allergy to 2-5 nuts
* Serum immunoglobulin E (IgE) >0.35 kilounits/L (kU/L) (determined by UniCAP within the past 12 months) and/or a SPT to nut >3 mm compared to control
* Positive oral food challenge (OFC) to less than 300mg of a nut in the nut mix at baseline (cumulative 444mg).

Exclusion Criteria:

* History of frequent or repeated, severe or life-threatening episodes of anaphylactic shock
* use of omalizumab or other non-traditional forms of allergen immunomodulatory therapy (not including corticosteroids) or biologic therapy in the 12 months prior to study entry
* history of eosinophilic gastrointestinal disease, uncontrolled asthma as defined by Global Initiative for Asthma (GINA)
* use of beta-blockers(oral)
* use of angiotensin-converting enzyme inhibitors (ACE)
* fails to tolerate 4mg of peanut after the first desensitization day
* Other significant medical conditions that in the opinion of the investigator prevent participation in the study,
* Previous intubation due to allergies or asthma,
* Symptomatic atopic dermatitis or chronic urticaria which may interfere with ability to evaluate oral immunotherapy and /or requiring daily medication including antihistamines,
* Patients with problems related to compliance or following study instructions, Inability to come to hospital every for dose escalation
* Pregnancy
* Non-fluency in English because participants may need to communicate with us after hours and be able to describe symptoms and concerns and follow instructions to treat anaphylaxis

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Desensitization to allergic food as assessed by change in maximum tolerated dose in a dichotomous manner | month 0, month 18
  Change in how much nuts the participant can eat without an allergic reaction after the low dose OIT assessed as dichotomous did the participant reach 5 times the baseline eliciting dose
Immunological change in IgG4 | month 0, month 18
  Change in allergen specific immunoglobulin G4 (IgG4) from baseline to end

SECONDARY OUTCOMES:
Desensitization to allergic food as assessed by change in maximum tolerated dose on a linear scale | month 0, month 18
  A continuous variable amount tolerated at baseline vs at end
Immunological change in IgG4 | pre-study, month 18
  Change in IgG4 from measures from historical data to 18 month of study. Some patients will have historical IgG4 values to compare
Desensitization to allergic food as assessed by maximum tolerated dose | month 18
  Did they reach 300mg (cumulative) on the 18 month exit oral food challenge
Desensitization to allergic food as assessed by maximum tolerated dose | month 0, month 18
  Did they reach 140mg (cumulative) on the 18 month exit oral food challenge

OTHER OUTCOMES:
Feasibility analysis as assessed by can the patients achieve the maintenance dosing of the allergen mix for OIT | month 18
  Proportion who achieve maintenance doses of their allergen mix (descriptive)
Feasibility analysis as assessed by drop-out rate | month 18
  Proportion who drop-out of the study (descriptive)
Incidence of Treatment-Emergent Adverse Events: Safety analysis as assessed by use of epinephrine | month 18
  Administration of epinephrine; (descriptive);
Quality of life scale | month 0, month 18
  Change in quality of life at 18m of children compared to baseline assessment (using validated questionnaire: Food allergy quality of life questionnaires (FAQLQ) FAQLQ Parental form (PF) for ages 0-12 OR the FAQLQ-teenager form (TF) using total score. The FAQLQ total and domain scores range from 1-7 with higher scores indicative of worse health related quality of life with the total score being the average of the domain scores. The domains include Emotional Impact, Social and Dietary Restrictions, Food Anxiety, Allergen Avoidance, and Risk of Accidental Exposure.
Change in allergen specific IgE, and components | month 0, month 18
  Change in allergen specific IgE, and components via microarray
Basophil activation test | month 0, month 18
  Basophil activation test
Skin prick test (SPT) reactivity to the individual nut extracts | month 0, month 18
  The size of the skin prick test will be compared
High content functional immune profiling via mass cytometry and single cell sorting | pre-study, month 18
  Compare the change in the immune pattern
Number of participants with treatment related adverse effects | month 0, month 18
  Diaries will be analyzed for allergic symptoms and tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Julia Upton, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03799328/Prot_SAP_000.pdf